CLINICAL TRIAL: NCT00087178
Title: A Clinical Trial Of Adjuvant Therapy Comparing Six Cycles Of 5-Fluorouracil, Epirubicin And Cyclophosphamide (FEC) To Four Cycles Of Adriamycin And Cyclophosphamide (AC) In Patients With Node-Negative Breast Cancer
Brief Title: Comparison of Two Combination Chemotherapy Regimens in Treating Women With Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP B-36; U10CA012027 (NIH)
Record Dates: First submitted 2004-07-08; First posted 2004-07-12 (Estimated); Results first posted 2022-08-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Doxorubicin; Epirubicin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1: adriamycin + cyclophosphamide (Active Comparator): Patients receive adriamycin IV over 15 minutes followed by cyclophosphamide IV over 30 minutes on day 1. Treatment repeats every 21 days for 4 courses.
  Interventions: Drug: cyclophosphamide; Drug: adriamycin
- Arm 2: fluorouracil + epirubicin + cyclophosphamide (Experimental): Patients receive fluorouracil IV, epirubicin IV over 15 minutes, and cyclophosphamide IV over 30 minutes on day 1. Treatment repeats every 21 days for 6 courses.
  Interventions: Drug: cyclophosphamide; Drug: epirubicin; Drug: fluorouracil

INTERVENTIONS:
Drug: cyclophosphamide — Arm 1: cyclophosphamide 600 mg/m2 IV every 21 days for 4 cycles; Arm 2: cyclophosphamide 500 mg/m2 IV every 21 days for 6 cycles
Drug: adriamycin — adriamycin 60 mg/m2 IV every 21 days for 4 cycles
  Other Names: doxorubicin; doxorubicin hydrochloride
  Arms: Arm 1: adriamycin + cyclophosphamide
Drug: epirubicin — epirubicin 100 mg/m2 IV every 21 days for 6 cycles
  Other Names: epirubicin hydrochloride
  Arms: Arm 2: fluorouracil + epirubicin + cyclophosphamide
Drug: fluorouracil — fluorouracil 500 mg/m2 IV every 21 days for 6 cycles
  Other Names: 5-fluorouracil; 5-FU
  Arms: Arm 2: fluorouracil + epirubicin + cyclophosphamide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fluorouracil, epirubicin, cyclophosphamide, and doxorubicin, work in different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which combination chemotherapy regimen is more effective in treating breast cancer.

PURPOSE: This randomized phase III trial is studying two combination chemotherapy regimens to compare how well they work in treating women who have undergone surgery for breast cancer that has not spread to the lymph nodes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare disease-free survival of women with node-negative breast cancer treated with adjuvant fluorouracil, epirubicin, and cyclophosphamide vs doxorubicin and cyclophosphamide.

Secondary

* Compare survival, recurrence-free interval, and distant recurrence-free interval in patients treated with these regimens.
* Compare adverse events in patients treated with these regimens.
* Compare quality of life, with regard to physical functioning, vitality, symptoms, and rates of post-chemotherapy amenorrhea, in premenopausal patients treated with these regimens.
* Determine the effect of induction of post-chemotherapy amenorrhea on disease-free survival in premenopausal patients treated with these regimens.
* Correlate post-chemotherapy amenorrhea and disease-free survival with hormone receptor status in premenopausal patients treated with these regimens.
* Correlate changes in left ventricular ejection fraction (LVEF) with self-reported physical functioning in patients treated with these regimens.
* Compare the efficacy of these regimens in patients with Human Epidermal Growth Factor Receptor 2 (HER2)/neu and/or topoisomerase-2-alpha gene amplification.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to hormone receptor status (estrogen receptor [ER] positive or progesterone receptor [PR] positive vs ER negative or PR negative) and type of prior surgery (lumpectomy vs total mastectomy). Patients are randomized to 1 of 2 treatment arms.

* Arm 1: Patients receive doxorubicin IV over 15 minutes followed by cyclophosphamide IV over 30 minutes on day 1. Treatment repeats every 21 days for 4 courses.
* Arm 2: Patients receive fluorouracil IV, epirubicin IV over 15 minutes, and cyclophosphamide IV over 30 minutes on day 1. Treatment repeats every 21 days for 6 courses.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

All patients with ER- or PR-positive tumors receive hormonal therapy daily beginning within 3-12 weeks after the completion of chemotherapy and continuing for at least 5 years.

All patients who have undergone prior lumpectomy undergo whole-breast radiotherapy beginning as soon as possible after the completion of chemotherapy. Patients who have undergone prior total mastectomy may undergo chest wall radiotherapy at the investigator's discretion. Patients assigned to the partial breast irradiation (PBI) group of protocol NSABP-B-39 undergo PBI according to protocol-specific guidelines.

Quality of life is assessed at baseline, on day 1 of course 4 of chemotherapy, and then every 6 months for 3 years.

Patients are followed every 6 months for up to 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 2,700 patients (1,350 per treatment arm) will be accrued for this study within 3.75 years.

ELIGIBILITY:
Eligibility

* Patients must be greater than or equal to 18 years of age.
* The patient must have a life expectancy of at least 10 years, excluding her diagnosis of breast cancer. (Comorbid conditions and performance status should be taken into consideration, but not the diagnosis of breast cancer.)
* The interval between the last surgery for breast cancer treatment (lumpectomy, mastectomy, sentinel lymph node biopsy, axillary surgery, or re-excision of lumpectomy margins) and randomization must be no more than 84 days.
* The tumor must be invasive adenocarcinoma on histologic examination. (Patients with tumors that are pure tubular or mucinous adenocarcinomas are not eligible.)
* The primary tumor must be T1-3 by clinical and pathologic evaluation.
* Lymph nodes obtained from all axillary staging procedures must be pN0 according to pathologic staging criteria of the 6th edition of the American Joint Committee on Cancer (AJCC) Cancer Staging Manual.
* Patients must have undergone axillary nodal staging procedures, for example sentinel node (SN) biopsy alone, SN biopsy followed by axillary sampling or completion dissection, or axillary node dissection to obtain lymph nodes for pathologic evaluation. If the patient has palpable nodes, axillary dissection is required.
* Patients must have an estrogen receptor (ER) analysis performed on the primary tumor prior to randomization. If ER is negative, then progesterone receptor (PgR) analysis must be performed. If ER is positive, PgR analysis is desired, but not mandatory. ("Marginal" or "borderline" results [i.e., those not definitively negative] will be considered positive regardless of the methodology used.)
* Patients must have had either a lumpectomy or total mastectomy.
* Patients must have no clinical or radiologic evidence of metastatic disease.
* Patients with skeletal pain are eligible for inclusion in the study if bone scan or roentgenological examination fail to disclose metastatic disease. Suspicious findings must be confirmed as benign by x-ray, MRI, or biopsy.
* The patient's menopausal status must be determined prior to randomization.

  * Pre- and postmenopausal women are eligible. The following criteria will be used to define postmenopausal:
  * a prior documented bilateral oophorectomy, or
  * a history of at least 12 months without spontaneous menstrual bleeding, or
  * age 55 or older with a prior hysterectomy or
  * age 54 or younger with a prior hysterectomy without oophorectomy (or in whom the status of the ovaries is unknown), with a documented follicle-stimulating hormone (FSH) level demonstrating confirmatory elevation in the lab's postmenopausal range.
  * Women failing to meet one of these criteria will be classified as premenopausal.
* At the time of randomization, the patient must have had the following: history and physical exam, EKG, and PA and lateral chest x-ray or chest CT within the past 3 months; bilateral mammogram within the past 6 months; and pelvic exam (for women who have a uterus and who will be receiving tamoxifen) within the past year.
* Within 3 months prior to entry, the patient must have a baseline LVEF measured by Multi Gated Acquisition (MUGA) scan or echocardiogram equal to or greater than the lower limit of normal for the facility performing the procedure.
* At the time of randomization:

  * The postoperative absolute granulocyte count (AGC) must be greater than or equal to 1500/mm3 (or greater than or equal to 1200/mm3 if, in the opinion of the investigator, this represents an ethnic or racial variant of normal).
  * Postoperative platelet count must be greater than or equal to 100,000/mm3. Significant underlying hematologic disorders must be excluded when the platelet count is above the ULN for the lab.
  * There must be postoperative evidence of adequate hepatic function, i.e.,
  * total bilirubin must be less than or equal to ULN for the lab unless the patient has a chronic Grade 1 bilirubin elevation (greater than ULN to 1.5 x ULN) due to Gilbert's disease or similar syndrome due to slow conjugation of bilirubin; and
  * alkaline phosphatase must be less than 2.5 x ULN for the lab; and
  * the aspartate transaminase (AST) [serum glutamic-oxaloacetic transaminase (SGOT)] must be less than or equal to 1.5 x ULN for the lab.
  * There must be postoperative evidence of normal renal function (serum creatinine less than or equal to ULN).
* Patients with a history of non-breast malignancies are eligible if they have been disease-free for 5 or more years prior to randomization and are deemed by their physician to be at low risk for recurrence. Patients with the following cancers are eligible if diagnosed and treated within the past 5 years: carcinoma in situ of the cervix, melanoma in situ, and basal cell and squamous cell carcinoma of the skin.
* Special conditions for eligibility of lumpectomy patients: radiation therapy and surgery Patients treated by lumpectomy followed by breast radiation therapy must meet all the eligibility criteria in addition to the following:

  * Generally, lumpectomy should be reserved for tumors less than 5 cm. However, at the investigator's discretion, patients treated with lumpectomy for tumors greater than or equal to 5 cm are eligible if eligibility criteria for lumpectomy are met.
  * The margins of the resected specimen must be histologically free of invasive tumor and DCIS as determined by the local pathologist. In patients in whom pathologic examination demonstrates tumor present at the line of resection, additional operative procedures may be performed to obtain clear margins. This is permissible even if axillary dissection has been performed. Patients in whom tumor is still present at the resected margin after re-excision(s) must undergo total mastectomy to be eligible.
  * This is a node-negative study, therefore irradiation of regional lymph nodes is prohibited in this trial.
  * Whole breast irradiation is required unless the patient is assigned to the partial breast irradiation group on NSABP B-39.
  * Postmastectomy chest wall irradiation at the investigator's discretion is permitted. However, this is a node-negative study; therefore irradiation of regional lymph nodes is prohibited in this trial.

Ineligibility

* Male patients are not eligible for this study.
* Pure tubular or mucinous adenocarcinomas.
* Bilateral malignancy (including DCIS) or a mass or mammographic abnormality in the opposite breast suspicious for malignancy unless there is biopsy proof that the mass is not malignant.
* Primary tumor staged as T4 for any reason.
* Suspicious palpable nodes in the ipsilateral or contralateral axilla or palpable supraclavicular or infraclavicular nodes. Patients with these conditions are considered ineligible unless there is biopsy evidence that these are not involved with tumor.
* Prior history of breast cancer, including DCIS (patients with a history of lobular carcinoma in situ [LCIS] are eligible).
* Treatment including radiation therapy, chemotherapy, biotherapy, and/or hormonal therapy administered for the currently diagnosed breast cancer prior to randomization. The only exceptions are:

  * Hormonal therapy, which may have been given for up to a total of 28 days anytime after diagnosis and before study entry. In such a case, hormonal therapy must stop at or before randomization and be re-started, if indicated, following chemotherapy.
  * If patient is enrolled in NSABP B-39 and randomized to Group 2, partial breast irradiation (PBI) may be completed prior to beginning treatment on NSABP B-36.
* Prior anthracycline therapy for any malignancy.
* Any sex hormonal therapy, e.g., birth control pills, ovarian hormonal replacement therapy, etc.. (These patients are eligible if this therapy is discontinued prior to randomization.)
* Therapy with any hormonal agents such as raloxifene (Evista®), tamoxifen, or other selective estrogen receptor modulators (SERMs), either for osteoporosis or breast cancer prevention. (Patients are eligible only if these medications are discontinued prior to randomization. With the exception of tamoxifen, these medications are not permitted while on the study.)
* Cardiac disease that would preclude the use of anthracyclines. This includes:

  * any documented myocardial infarction;
  * angina pectoris that requires the use of anti-anginal medication;
  * any history of documented congestive heart failure;
  * serious cardiac arrhythmia requiring medication,
  * severe conduction abnormality;
  * valvular disease with documented cardiac function compromise; and
  * poorly controlled hypertension, i.e., diastolic greater than 100 mm/Hg. (Patients with hypertension that is well controlled on medication are eligible for entry.)
* Non-malignant systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude a patient from being subjected to any of the treatment options or would prevent prolonged follow-up.
* Pregnancy or lactation at the time of proposed randomization. Women of reproductive potential must agree to use an effective non-hormonal method of contraception.
* Concurrent treatment with investigational agents.
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements.
* Special conditions for ineligibility of lumpectomy patients: radiation therapy and surgery. For patients treated by lumpectomy, breast irradiation is required. The following patients will be ineligible:

  * Patients with diffuse tumors (as demonstrated on mammography) that would not be considered surgically amenable to lumpectomy. (These patients are eligible if they undergo mastectomy.)
  * Patients treated with lumpectomy in whom there is another clinically dominant mass or mammographically suspicious abnormality within the ipsilateral breast remnant. Such a mass must be biopsied and demonstrated to be histologically benign prior to randomization or, if malignant, must be surgically removed with clear margins.
  * Patients in whom the margins of the resected specimen are involved with invasive tumor or ductal carcinoma in situ (DCIS). Additional surgical resections to obtain free margins are allowed. Patients in whom tumor is still present after the additional resection(s) must undergo mastectomy to be eligible. (Patients with margins positive for LCIS are eligible without additional resection.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2722 (Actual)
Dates: Start 2004-05; Primary Completion 2014-03 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman Wolmark, MD, Principal Investigator — NSABP Foundation Inc
Locations (606):
- United States (586):
  - Clearview Cancer Institute, Huntsville, Alabama
  - Providence Cancer Center, Anchorage, Alaska
  - Banner Thunderbird Medical Center, Glendale, Arizona
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - CCOP - Western Regional, Arizona, Phoenix, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Alta Bates Summit Comprehensive Cancer Center, Berkeley, California
  - Peninsula Medical Center, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - North Bay Cancer Center, Fairfield, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Valley Medical Oncology, Fremont, California
  - Glendale Memorial Hospital Comprehensive Cancer Center, Glendale, California
  - California Cancer Care, Incorporated - Greenbrae, Greenbrae, California
  - Marin Cancer Institute at Marin General Hospital, Greenbrae, California
  - Sutter Health - Western Division Cancer Research Group, Greenbrae, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Scripps Cancer Center - San Diego, La Jolla, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Pacific Shores Medical Group - Long Beach, Long Beach, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Chao Family Comprehensive Cancer Center at University of California Irvine Medical Center, Orange, California
  - Valley Care Medical Center, Pleasanton, California
  - Valley Medical Oncology Consultants - Pleasanton, Pleasanton, California
  - North Valley Breast Clinic, Redding, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - Sutter Cancer Center at Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Office -Vandever Medical Office, San Diego, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Cancer Center of Santa Barbara, Santa Barbara, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Stanford Cancer Center, Stanford, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Sutter Solano Medical Center, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Poudre Valley Hospital, Fort Collins, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Helen and Harry Gray Cancer Center at Hartford Hospital, Hartford, Connecticut
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Kent General Hospital, Dover, Delaware
  - Tunnell Cancer Center at Beebe Medical Center, Lewes, Delaware
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Lombardi Comprehensive Cancer Center at Georgetown University Medical Center, Washington D.C., District of Columbia
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Morton Plant Hospital, Clearwater, Florida
  - Herbert D. Kerman Regional Oncology Center - Daytona Beach, Daytona Beach, Florida
  - Michael and Dianne Bienes Comprehensive Cancer Center at Holy Cross Hospital, Fort Lauderdale, Florida
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Ella Milbank Foshay Cancer Center at Jupiter Medical Center, Jupiter, Florida
  - Center for Cancer Care and Research at Watson Clinic, LLP, Lakeland, Florida
  - Lakeland Regional Cancer Center at Lakeland Regional Medical Center, Lakeland, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - Piedmont Hospital, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Augusta Oncology Associates - Walton Way, Augusta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Curtis and Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - St. Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Sherman Hospital, Elgin, Illinois
  - Alexian Brothers Radiation Oncology, Elk Grove Village, Illinois
  - Eureka Community Hospital, Eureka, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Galesburg Clinic, PC, Galesburg, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Delnor Community Hospital - Geneva, Geneva, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Hopedale Medical Complex, Hopedale, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - Provena St. Mary's Regional Cancer Center - Kankakee, Kankakee, Illinois
  - La Grange Memorial Hospital, La Grange, Illinois
  - McDonough District Hospital, Macomb, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - BroMenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center, Normal, Illinois
  - Saint James Hospital and Health Centers Comprehensive Cancer Institute - Olympia Fields, Olympia Fields, Illinois
  - Community Hospital of Ottawa, Ottawa, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Ottawa, Ottawa, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Cancer Treatment Center at Pekin Hospital, Pekin, Illinois
  - Proctor Hospital, Peoria, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Oncology Hematology Associates of Central Illinois, PC - Peoria, Peoria, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - OSF St. Francis Medical Center, Peoria, Illinois
  - Illinois Valley Community Hospital, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Center for Cancer Care at OSF Saint Anthony Medical Center, Rockford, Illinois
  - St. Margaret's Hospital, Spring Valley, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Francis Hospital and Health Centers - Beech Grove Campus, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology, Fort Wayne, Indiana
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Clarian Arnett Cancer Care, Lafayette, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - Community Hospital, Munster, Indiana
  - Reid Hospital & Health Care Services, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Covenant Cancer Treatment Center, Waterloo, Iowa
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - Providence Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Johnson County Radiation Therapy, Overland Park, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Shawnee Mission Medical Center, Shawnee Mission, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Cancer Resource Center at King's Daughters Medical Center, Ashland, Kentucky
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Louisville Oncology at Norton Cancer Institute - Louisville, Louisville, Kentucky
  - Baptist Hospital East - Louisville, Louisville, Kentucky
  - Pennington Cancer Center at Baton Rouge General, Baton Rouge, Louisiana
  - Ochsner Health Center - Bluebonnet, Baton Rouge, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Drs Gurtler Brinz and Russo APMC-Metairie Oncologists, Metairie, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Ochsner Cancer Institute at Ochsner Clinic Foundation, New Orleans, Louisiana
  - Christus Schumpert Cancer Treatment Center, Shreveport, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Harbor View Cancer Center at Harbor Hospital, Baltimore, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Harry & Jeanette Weinberg Cancer Institute at Franklin Square Hospital Center, Baltimore, Maryland
  - Suburban Hospital, Bethesda, Maryland
  - Union Hospital Cancer Program at Union Hospital, Elkton, Maryland
  - Kaiser Permanente Mid-Atlantic Medical Group-Largo Medical Facility, Largo, Maryland
  - St. Mary's Hospital, Leonardtown, Maryland
  - Kaiser Permanente - Towson, Lutherville, Maryland
  - Kaiser Permanente Capital Area Medical Group - Shady Grove Facility, Rockville, Maryland
  - Peninsula Regional Medical Center, Salisbury, Maryland
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Commonwealth Hematology-Oncology, PC - Concord, Concord, Massachusetts
  - Commonwealth Hematology Oncology PC - Dorchester, Dorchester, Massachusetts
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - Commonwealth Hematology-Oncology, PC - Haverhill, Haverhill, Massachusetts
  - Commonwealth Hematology-Oncology, PC - Lawrence, Lawrence, Massachusetts
  - Commonwealth Hematology Oncology PC - Leominster, Leominster, Massachusetts
  - Commonwealth Hematology Oncology PC - Milton, Milton, Massachusetts
  - Berkshire Hematology Oncology, PC, Pittsfield, Massachusetts
  - Jordan Hospital Club Cancer Center, Plymouth, Massachusetts
  - Commonwealth Hematology-Oncology, PC - Quincy, Quincy, Massachusetts
  - Commonwealth Hematology-Oncology, PC - Stoneham, Stoneham, Massachusetts
  - Commonwealth Hematology-Oncology, PC - Weymouth, Weymouth, Massachusetts
  - Commonwealth Hematology-Oncology, PC - Worcester, Worcester, Massachusetts
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County Medical Center, Big Rapids, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Great Lakes Cancer Institute at McLaren Regional Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Health Care, Grand Rapids, Michigan
  - Metro Health Hospital, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Lapeer Regional Hospital, Lapeer, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - Upper Michigan Cancer Center at Marquette General Hospital, Marquette, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - Oncology Care Associates, PLLC, Saint Joseph, Michigan
  - Providence Cancer Institute at Providence Hospital - Southfield Campus, Southfield, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Hattiesburg Clinic, PA at Forrest General, Hattiesburg, Mississippi
  - Hematology & Oncology Clinic, Hattiesburg, Mississippi
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Saint Luke's Hospital, Chesterfield, Missouri
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Independence Regional Health Center, Independence, Missouri
  - Freeman Cancer Institute at Freeman Health System, Joplin, Missouri
  - St. John's Regional Medical Center, Joplin, Missouri
  - Truman Medical Center - Hospital Hill, Kansas City, Missouri
  - Saint Luke's Cancer Institute at Saint Luke's Hospital, Kansas City, Missouri
  - Kansas City Cancer Center at St. Joseph's Medical Mall, Kansas City, Missouri
  - St. Joseph Medical Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Parvin Radiation Oncology, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - Radiation Oncology Associates of Kansas City at Northland Radiation Oncology Center, Kansas City, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Midwest Hematology Oncology Group, Incorporated, St Louis, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - Arch Medical Services, Incorporated at Center for Cancer Care and Research, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Renown Institute for Cancer at Renown Regional Medical Center, Reno, Nevada
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Mountainside Hospital Cancer Center, Montclair, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Warren Hospital, Phillipsburg, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Hematology Oncology Associates, PC, Albuquerque, New Mexico
  - Lovelace Medical Center - Gibson, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - New York Oncology Hematology, PC at Albany Regional Cancer Care, Albany, New York
  - New York Oncology Hematology, PC at Albany Medical Center, Albany, New York
  - Amsterdam Community Cancer Program, Amsterdam, New York
  - Finger Lakes Hematology and Oncology, Clifton Springs, New York
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - Charles R. Wood Cancer Center at Glens Falls Hospital, Glens Falls, New York
  - New York Oncology Hematology, PC - Hudson, Hudson, New York
  - Queens Cancer Center of Queens Hospital, Jamaica, New York
  - New York Oncology Hematology, PC - Latham, Latham, New York
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Don Monti Comprehensive Cancer Center at North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Riverview Cancer Care Medical Associates, PC, Rexford, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Samaritan Hospital at Northeast Health, Troy, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Alamance Cancer Center at Alamance Regional Medical Center, Burlington, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - John Smith, Jr. - Dalton McMichael Cancer Center at Morehead Memorial Hospital, Eden, North Carolina
  - Cape Fear Valley Medical Center Cancer Center, Fayetteville, North Carolina
  - CaroMont Cancer Center at Gaston Memorial Hospital, Gastonia, North Carolina
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Leo W. Jenkins Cancer Center at ECU Medical School, Greenville, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Marion L. Shepard Cancer Center at Beaufort County Hospital, Washington, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Medcenter One Hospital Cancer Care Center, Bismarck, North Dakota
  - Mid Dakota Clinic, PC, Bismarck, North Dakota
  - St. Alexius Medical Center Cancer Center, Bismarck, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - MeritCare Broadway, Fargo, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Christ Hospital Cancer Center, Cincinnati, Ohio
  - Oncology Hematology Care, Incorporated - Blue Ash, Cincinnati, Ohio
  - Charles M. Barrett Cancer Center at University Hospital, Cincinnati, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Middletown Regional Hospital, Franklin, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - United States Air Force Medical Center - Wright-Patterson, Wright-Patterson Air Force Base, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Tod Children's Hospital, Youngstown, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Cleo Craig Cancer Research Clinic, Lawton, Oklahoma
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Cancer Care Associates - Mercy Campus, Oklahoma City, Oklahoma
  - LaFortune Cancer Center at St. John Medical Center, Tulsa, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Kaiser Permanente Health Care - Portland, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, PC at Hahne Regional Cancer Center, DuBois, Pennsylvania
  - Dale and Frances Hughes Cancer Center at Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Easton Regional Cancer Center at Easton Hospital, Easton, Pennsylvania
  - Ephrata Cancer Center at Ephrata Community Hospital, Ephrata, Pennsylvania
  - Regional Cancer Center - Erie, Erie, Pennsylvania
  - Saint Vincent Health Center, Erie, Pennsylvania
  - PinnacleHealth Regional Cancer Center at Polyclinic Hospital, Harrisburg, Pennsylvania
  - Richard G. Laube Cancer Center at ACMH, Kittanning, Pennsylvania
  - Riddle Memorial Hospital Cancer Center, Media, Pennsylvania
  - Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Frankford Hospital Cancer Center - Torresdale Campus, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Western Pennsylvania Cancer Institute at Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Guthrie Cancer Center at Guthrie Clinic Sayre, Sayre, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates of Northeastern Pennsylvania, Scranton, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Associates in Hematology-Oncology, PC at Crozer Regional Cancer Center, Upland, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - Hematology and Oncology Associates of Rhode Island, Cranston, Rhode Island
  - Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - Kent County Memorial Hospital, Warwick, Rhode Island
  - AnMed Cancer Center, Anderson, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Oncology Services of Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - U.T. Medical Center Cancer Institute, Knoxville, Tennessee
  - Texas Oncology - Midtown Austin, Austin, Texas
  - Texas Oncology, PA at Texas Oncology Cancer Center - Central, Austin, Texas
  - Texas Oncology, PA at South Austin Cancer Center, Austin, Texas
  - St. Joseph Regional Cancer Center, Bryan, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - Texas Oncology, PA at Texas Cancer Center Round Rock, Round Rock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Green Mountain Oncology Group, Bennington, Vermont
  - Kaiser Permanente Medical Center - Fair Oaks, Fairfax, Virginia
  - Virginia Oncology Associates - Hampton, Hampton, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Virginia Cancer Institute - West End, Richmond, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Carilion Cancer Center of Western Virginia, Roanoke, Virginia
  - Overlake Cancer Center at Overlake Hospital Medical Center, Bellevue, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Rockwood Clinic Cancer Treatment Center, Spokane, Washington
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - Providence Cancer Center at Holy Family Hospital, Spokane, Washington
  - Cancer Care Northwest - North, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - St. Mary Regional Cancer Center at St. Mary Medical Center, Walla Walla, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - Edwards Comprehensive Cancer Center at Cabell Huntington Hospital, Huntington, West Virginia
  - St. Mary's Regional Cancer Center at St. Mary's Medical Center, Huntington, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Princeton Community Hospital, Princeton, West Virginia
  - Center for Cancer Treatment & Prevention at Sacred Heart Hospital, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Care at Regional Cancer Center, Eau Claire, Wisconsin
  - Vince Lombardi Cancer Center at Aurora Lakeland Medical Center - Elkhorn, Elkhorn, Wisconsin
  - Central Wisconsin Cancer Program at Agnesian HealthCare, Fond du Lac, Wisconsin
  - Oncology Alliance, SC - Milwaukee - East, Glendale, Wisconsin
  - Green Bay Oncology, Limited at St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Dean Medical Center - Madison, Madison, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Medical Consultants, Limited, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Marshfield Clinic - Lakeland Center, Minocqua, Wisconsin
  - Ministry Medical Group at Saint Mary's Hospital, Rhinelander, Wisconsin
  - Marshfield Clinic - Indianhead Center, Rice Lake, Wisconsin
  - Saint Michael's Hospital Cancer Center, Stevens Point, Wisconsin
  - Vince Lombardi Cancer Clinic - Two Rivers, Two Rivers, Wisconsin
  - Marshfield Clinic - Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming
- Canada (16):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Trillium Health Centre - Mississauga Site, Mississauga, Ontario
  - Carlo Fidani Peel Regional Cancer Centre at Credit Valley Hospital, Mississauga, Ontario
  - Ottawa Hospital Regional Cancer Centre - General Campus, Ottawa, Ontario
  - Edmond Odette Cancer Centre at Sunnybrook, Toronto, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - CHUM - Hotel Dieu Hospital, Montreal, Quebec
  - CHUM - Hopital Saint-Luc, Montreal, Quebec
  - Royal Victoria Hospital - Montreal, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital - Montreal, Montreal, Quebec
  - Hopital du Saint-Sacrement - Quebec, Québec, Quebec
- Puerto Rico (4):
  - Andres Grillasca Hospital, Ponce
  - Hato Rey Hematology/Oncology Group, PSC, San Juan
  - I. Gonzalez Martinez Oncologic Hospital, San Juan
  - San Juan City Hospital, San Juan

REFERENCES:
- [Derived] Geyer CE Jr, Bandos H, Rastogi P, Jacobs SA, Robidoux A, Fehrenbacher L, Ward PJ, Polikoff J, Brufsky AM, Provencher L, Paterson AHG, Hamm JT, Carolla RL, Baez-Diaz L, Julian TB, Swain SM, Mamounas EP, Wolmark N. Definitive results of a phase III adjuvant trial comparing six cycles of FEC-100 to four cycles of AC in women with operable node-negative breast cancer: the NSABP B-36 trial (NRG Oncology). Breast Cancer Res Treat. 2022 Jun;193(3):555-564. doi: 10.1007/s10549-021-06417-y. Epub 2022 Mar 1. PMID 35230585
- [Derived] Ganz PA, Bandos H, Geyer CE Jr, Robidoux A, Paterson AHG, Polikoff J, Baez-Diaz L, Brufsky AM, Fehrenbacher L, Parsons AW, Ward PJ, Provencher L, Hamm JT, Stella PJ, Carolla RL, Margolese RG, Shibata HR, Perez EA, Wolmark N. Behavioral and health outcomes from the NRG Oncology/NSABP B-36 trial comparing two different adjuvant therapy regimens for early-stage node-negative breast cancer. Breast Cancer Res Treat. 2022 Feb;192(1):153-161. doi: 10.1007/s10549-021-06475-2. Epub 2022 Feb 3. PMID 35112166

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm 1: Adriamycin + Cyclophosphamide | Arm 2: Fluorouracil + Epirubicin + Cyclophosphamide
Started | 1361 | 1361
Completed | 1355 | 1343
Not Completed | 6 | 18
Not completed — No follow up data | 5 | 15
Not completed — No clinical assessment | 1 | 2
Not completed — Patient not at risk for primary endpoint | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 1- Adriamycin + Cyclophosphamide: Patients receive adriamycin IV over 15 minutes followed by cyclophosphamide IV over 30 minutes on day 1. Treatment repeats every 21 days for 4 courses.
  cyclophosphamide: Arm 1:cyclophosphamide 600 mg/m2 IV every 21 days for 4 cycles; Arm 2: cyclophosphamide 500 mg/m2 IV every 21 days for 6 cycles
  adriamycin: adriamycin 60 mg/m2 IV every 21 days for 4 cycles
- Arm 2 - Fluorouracil + Epirubicin + Cyclophosphamide: Patients receive fluorouracil IV, epirubican IV over 15 minutes, and cyclophosphamide IV over 30 minutes on day 1. Treatment repeats every 21 days for 6 courses.
  cyclophosphamide: Arm 1: cyclophosphamide 600 mg/m2 IV every 21 days for 4 cycles; Arm 2: cyclophosphamide 500 mg/m2 IV every 21 days for 6 cycles
  epirubicin: epirubicin 100 mg/m2 IV every 21 days for 6 cycles
  fluorouracil: fluorouracil 500 mg/m2 IV every 21 days for 6 cycles
- Total: Total of all reporting groups
Arm/Group | Arm 1- Adriamycin + Cyclophosphamide | Arm 2 - Fluorouracil + Epirubicin + Cyclophosphamide | Total
Number analyzed (Participants) | 1361 | 1361 | 2722
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (9.4) | 52 (9.6) | 52 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1361 | 1361 | 2722
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival
Description: Percentage of patients free from DFS event. DFS events include local, regional, or distant recurrence, second primary cancer or death from any cause prior to recurrence or second primary cancer
Time Frame: 9 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Adriamycin + Cyclophosphamide | Arm 2: Fluorouracil + Epirubicin + Cyclophosphamide
Number analyzed (Participants) | 1355 | 1343
percentage of participants | 80.1 | 79.4

2. Secondary Outcome: Survival
Description: Percentage of patients alive
Time Frame: 9 years
Population: Patients with any type of follow-up.
Measure: Number; unit: percentage of participants alive
Arm/Group | Arm 1: Adriamycin + Cyclophosphamide | Arm 2: Fluorouracil + Epirubicin + Cyclophosphamide
Number analyzed (Participants) | 1356 | 1345
percentage of participants alive | 89.8 | 89.9

3. Secondary Outcome: Adverse Events
Description: Percentage of patients with at least one grade 2 or higher adverse event reported
Time Frame: 9 years
Population: Patients with follow-up and available adverse event information.
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Adriamycin + Cyclophosphamide | Arm 2: Fluorouracil + Epirubicin + Cyclophosphamide
Number analyzed (Participants) | 1349 | 1333
percentage of participants | 28.5 | 45.0

4. Secondary Outcome: Quality of Life-Functional Assessment of Cancer Therapy
Description: Functional Assessment of Cancer Therapy (FACT-B) trial outcome index (TOI) score. FACT-B TOI score ranges from 0 to 92, with a higher score indicating better QOL.
Time Frame: 12 months
Population: Patients who participated in the QOL sub-study
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm 1: Adriamycin + Cyclophosphamide | Arm 2: Fluorouracil + Epirubicin + Cyclophosphamide
Number analyzed (Participants) | 675 | 656
score on a scale
  Score day 1 cycle 4 | 61.7 [60.9 to 62.7] | 60.3 [59.4 to 61.2]
  Score 6 months | 69.2 [68.3 to 70.1] | 66.9 [66.0 to 67.8]
  Score 12 months | 71.7 [70.8 to 72.7] | 71.1 [70.2 to 72.0]

5. Secondary Outcome: Post Chemotherapy Amenorrhea
Description: Percent with post chemotherapy amenorrhea
Time Frame: 18 months
Population: Patients who participated in the Menstrual History sub-study
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Adriamycin + Cyclophosphamide | Arm 2: Fluorouracil + Epirubicin + Cyclophosphamide
Number analyzed (Participants) | 474 | 451
percentage of participants | 59.1 | 67.4

6. Secondary Outcome: Change in Left Ventricular Ejection Fraction (LVEF) at the 12-month Evaluation
Description: Change in LVEF from randomization to 12 months
Time Frame: 12 months
Population: Patients who participated in the cardiac function sub-study
Measure: Mean (95% Confidence Interval); unit: Change in percent ejection fraction
Arm/Group | Arm 1: Adriamycin + Cyclophosphamide | Arm 2: Fluorouracil + Epirubicin + Cyclophosphamide
Number analyzed (Participants) | 159 | 146
Change in percent ejection fraction | -2.61 [-3.70 to -1.53] | -2.65 [-3.79 to -1.52]

7. Secondary Outcome: HER-2 and Topo II Gene Amplification
Time Frame: 6 years
Population: Data were not collected. Gene amplification analysis was not performed on the submitted blocks.
Arm/Group | Arm 1: Adriamycin + Cyclophosphamide | Arm 2: Fluorouracil + Epirubicin + Cyclophosphamide
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Recurrence-free Interval
Description: Percentage of patients with local-regional recurrence or distant recurrence
Time Frame: 9 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Adriamycin + Cyclophosphamide | Arm 2: Fluorouracil + Epirubicin + Cyclophosphamide
Number analyzed (Participants) | 1355 | 1343
percentage of participants | 10.8 | 10.4

9. Secondary Outcome: Distant Recurrence-free Interval
Description: Percentage of patients with distant recurrence
Time Frame: 9 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1: Adriamycin + Cyclophosphamide | Arm 2: Fluorouracil + Epirubicin + Cyclophosphamide
Number analyzed (Participants) | 1355 | 1343
percentage of participants | 8.3 | 7.2

ADVERSE EVENTS:
Description: Participants at Risk includes any patient who submitted an AE form.
Groups:
- Adriamycin + Cyclophosphamide: Patients receive adriamycin IV over 15 minutes followed by cyclophosphamide IV over 30 minutes on day 1. Treatment repeats every 21 days for 4 courses.
  cyclophosphamide: Arm 1: cyclophosphamide 600 mg/m2 IV every 21 days for 4 cycles; Arm 2: cyclophosphamide 500 mg/m2 IV every 21 days for 6 cycles
  adriamycin: adriamycin 60 mg/m2 IV every 21 days for 4 cycles
- Fluorouracil + Epirubicin + Cyclophosphamide: Patients receive fluorouracil IV, epirubicin IV over 15 minutes, and cyclophosphamide IV over 30 minutes on day 1. Treatment repeats every 21 days for 6 courses.
  cyclophosphamide: Arm 1: cyclophosphamide 600 mg/m2 IV every 21 days for 4 cycles; Arm 2: cyclophosphamide 500 mg/m2 IV every 21 days for 6 cycles
  epirubicin: epirubicin 100 mg/m2 IV every 21 days for 6 cycles
  fluorouracil: fluorouracil 500 mg/m2 IV every 21 days for 6 cycles
Arm/Group | Adriamycin + Cyclophosphamide | Fluorouracil + Epirubicin + Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 12/1351 | 26/1337
Other Adverse Events (participants affected / at risk) | 290/1351 | 454/1337
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adriamycin + Cyclophosphamide (N=1351) | Fluorouracil + Epirubicin + Cyclophosphamide (N=1337)
Agitation (Psychiatric disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Colonic perforation (Gastrointestinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Heart failure (Cardiac disorders) | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 1 | 2
Pericardial effusion (Cardiac disorders) | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 1
Platelet count decreased (Investigations) | 3 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Stroke (Nervous system disorders) | 0 | 2
Sudden death NOS (General disorders) | 1 | 2
Syncope (Nervous system disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 4
Uterine hemorrhage (Reproductive system and breast disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Leukemia secondary to oncology chemotherapy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
White blood cell decreased (Investigations) | 0 | 1
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Enterocolitis infectious (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adriamycin + Cyclophosphamide (N=1351) | Fluorouracil + Epirubicin + Cyclophosphamide (N=1337)
Anemia (Blood and lymphatic system disorders) | 106 | 147
Fatigue (General disorders) | 118 | 165
Febrile neutropenia (Blood and lymphatic system disorders) | 50 | 127
Mucositis oral (Gastrointestinal disorders) | 42 | 81
Nausea (Gastrointestinal disorders) | 94 | 121
Neutrophil count decreased (Investigations) | 80 | 92
Platelet count decreased (Investigations) | 25 | 84
Vomiting (Gastrointestinal disorders) | 62 | 99

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less